CLINICAL TRIAL: NCT00775710
Title: A Randomized Controlled Trial Comparing Two Protocols to Withdraw Non-invasive Ventilation (NIV) After an Episode of Hypercapnic Respiratory Failure
Brief Title: Clinical Trial Assessing Two Protocols to Withdraw Non-invasive Ventilation in Hypercapnic Respiratory Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Dr. Jacobo Sellares, Respiratoy Intensive Care Unit
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NIV-JS1
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2008-10

CONDITIONS: Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Non-invasive ventilation is maintained during three nights after recovery of an episode of hypercapnic respiratory failure.
  Interventions: Device: Nocturnal non-invasive ventilation
- 2 (No Intervention): Discontinuation of NIV after the recovery of hypercapnic respiratory failure, without prolong it during night.

INTERVENTIONS:
Device: Nocturnal non-invasive ventilation — Prolongation of non-invasive ventilation during 3 nights.
  Arms: 1

SUMMARY:
The purpose of the study is to determine the optimal method to withdraw non-invasive ventilation after an episode of hypercapnic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Acute hypercapnic respiratory failure.
* Use of NIV to treat respiratory failure.
* Persistence of hypercapnia after discontinuation of NIV

Exclusion Criteria:

* Home NIV
* Facial or cranial trauma or surgery,
* Recent gastric or esophageal surgery,
* Active upper gastrointestinal bleeding,
* Excessive amount of respiratory secretions,
* Tracheostomy
* Lack of cooperation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2006-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
New episode of hypercapnic respiratory failure after discontinuation of non-invasive ventilation | At the end of enrollment time

SECONDARY OUTCOMES:
Incidence of long term dependency on non-invasive ventilation | At the end of enrollment time
Hospital and 6-month survival | At the end of enrollment time

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Sellares, MD, Principal Investigator — Hospital Clinic
Locations (3):
- Spain (3):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona

REFERENCES:
- [Derived] Sellares J, Ferrer M, Anton A, Loureiro H, Bencosme C, Alonso R, Martinez-Olondris P, Sayas J, Penacoba P, Torres A. Discontinuing noninvasive ventilation in severe chronic obstructive pulmonary disease exacerbations: a randomised controlled trial. Eur Respir J. 2017 Jul 5;50(1):1601448. doi: 10.1183/13993003.01448-2016. Print 2017 Jul. PMID 28679605